CLINICAL TRIAL: NCT06832059
Title: Precision Nutrition Versus Standard Dietary Care: Continuous Glucose Monitoring as a Tool for Guided Nutrition Care in Type 2 Diabetes - The PRECISE-DIET Trial. -A Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Bettina Ewers, Head of Nutrition and PhD, Steno Diabetes Center Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-24083559
Record Dates: First submitted 2025-01-09; First posted 2025-02-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Dietary intervention; CGM; continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Precise diet intervention (Experimental): The precise diet intervention for 12 weeks (n=20).
  Interventions: Other: The precise diet intervention

INTERVENTIONS:
Other: The precise diet intervention — The intervention includes training and education in CGM use and reduction in overall carbohydrate intake guided by individualized flexible nutrition recommendations, with adjustments made according to postprandial blood glucose responses. Staff will guide participants in the daily carbohydrate intake with personalized adjustments to accommodate individual needs by the individuals. The primary goal is to minimize the participant's time spent above 10 mmol/l

SUMMARY:
The primary aim of this pilot study is to assess the feasibility of a 12-week dietary intervention combined with the use of CGM in adults with T2D. The results of the pilot study will provide insights into recruitment, design, and the effectiveness of the intervention for the future long-term (12-month) PRECISE-DIET STUDY

DETAILED DESCRIPTION:
In recent decades, there has been a significant rise in the development and use of glucose lowering drugs aimed at improving glycemic control in individuals with type 2 diabetes (T2D). Despite medical advancements, more than one-third of the danish population with T2D have a hemoglobin A1c (HbA1c) exceeding the recommended thresholds. One limiting factor in supporting individuals achieve their glycaemic target may be driven by substantial postprandial increases in plasma glucose levels, which is influenced by the quantity and type of carbohydrates in meals, underscoring the critical role of dietary interventions as an integral component of T2D management.

Recent studies have demonstrated that the use of continuous glucose monitors (CGMs), which allow individuals to track their glucose profiles continuously throughout the day, improves glycemic control in T2D patients. However, these studies often exclude dietary interventions, which could potentially yield greater improvements in blood glucose regulation.

Nutritional research in recent years has focused on dietary patterns such as low-fat diets, the paleo diet, and vegan diets. Nevertheless, these studies have not sufficiently addressed individualized dietary adjustments to mitigate postprandial glucose excursions, despite their substantial importance for glycemic control.

Several clinical studies have revealed significant inter-individual variations in glycemic responses to identical standardized meals, highlighting the necessity of a personalized approach to dietary recommendations, particularly with a focus on carbohydrate intake.

The primary aim of this pilot study is to assess the feasibility of a 12-week dietary intervention combined with the use of CGM in adults with T2D. The results of the pilot study will provide insights into recruitment, design, and the effectiveness of the intervention for the future long-term (12-month) PRECISE-DIET STUDY

ELIGIBILITY:
Inclusion Criteria:

* T2D

  * Diabetes duration of ≥12 months
  * ≥18 years of age
  * HbA1c ≥58 mmol/mol
  * Attending the SDCC outpatient clinic
  * Provided voluntary signed informed consent.

Exclusion Criteria:

* Inability to understand the patient information.
* Complications which do not permit to lowering HbA1c to <58 mmol/mol.
* Treatment with insulin.
* Low daily carbohydrate intake (defined as below 25 E% or 100 g/day) prior to study inclusion.
* Systematic use of corticosteroids.
* Using or requiring a specialized diet (e.g., kidney diet).
* Circumstances that affect HbA1c (e.g., liver disease and anaemia).
* Known or suspected drug or alcohol abuse (judged by the investigator).
* Pregnancy or breastfeeding or plans of pregnancy within the study period.
* Participation in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Fidelity testing | 12 weeks after baseline
  Participants will be invited to a workshop to evaluate the intervention and its components. Procedures from fidelity testing will be applied in the evaluation. These specific topics will be evaluated:
  * Study design
    o Is the design appropriate? E.g., number of visits, CGM use, dietetic feedback?
  * Sampling strategy
    o E.g., how many participated, recruitment methods, sample diversity?
  * Treatment receipt
    * "What is learned?"
    * Is the intervention relevant to and accepted by the participants?
  * Treatment enactment
    * What is actually used and done?
    * Do participants' "behavioural skills" improve?

SECONDARY OUTCOMES:
HbA1c (mmol/mol) | Measured at baseline and after 12 weeks
  Assessed from blood samples
Time in range (TIR) | Measured at baseline and after 12 weeks
  Time spent in time in range 3.9 mmol/l - 10.0 mmol/l from CGM data
Time above range (TAR) | Measured at baseline and after 12 weeks
  Time spent in time above range 10.1-13.9 mmol/l from CGM data
Time below range (TBR) | Measured at baseline and after 12 weeks
  Time spent in time below range <3.9 mmol/l from from CGM data
Coefficient of variation (CV) | Measured at baseline and after 12 weeks
  Percentage coefficient of variation in glucose differences
Estimated HbA1c | Measured at baseline and after 12 weeks
  Estimated HbA1c (14-days average of the CGM data)
Body mass index (kg/m^2) | Measured at baseline and after 12 weeks
  Calculated from body weight (kg) and height (m).
Body weight (kg) | Measured at baseline and after 12 weeks
  Measured on a digital scale
Waist circumference (cm) | Measured at baseline and after 12 weeks
  Measured using tape measure.
Hip circumference (cm) | Measured at baseline and after 12 weeks
  Measured using tape measure
Systolic blood pressure (mmHg) | Measured at baseline and after 12 weeks
  Measured under resting
Diastolic blood pressure (mmHg) | Measured at baseline and after 12 weeks
  Measured under resting
Self-reported diabetes distress | Measured at baseline and after 12 weeks
  Assessed from the Problem Areas in Diabetes Scale comprising of twenty emotional-distress questions. Each item can be rated from 0 to 5.
Self-reported treatment satisfaction | Measured at baseline and after 12 weeks
  Assessed from the questionnaire Diabetes Treatment Satisfaction Questionnaire (DTSQ).
Dietary intake | Measured at baseline and after 12 weeks
  Dietary intake (total energy intake and macronutrient composition based on 3-days' diet records)

OTHER OUTCOMES:
Changes in glucose lowering drugs | Measured at baseline and after 12 weeks
  Medication status, change in doses or discontinuation of medicine
Personality trait assesment | Baseline
  Assesed fromt the BIG FIVE Inventory questionnaire (BFI-44). Comprising of 44 items.
Physical activity | Measured at baseline and after 12 weeks
  Physical activity levels measured by X3 accelerometers

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Ewers, PhD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No